CLINICAL TRIAL: NCT00978198
Title: ASP1517 Phase 1 Clinical Study - Single and Multiple Oral Dosing of ASP1517 in Healthy Non-elderly Male Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetic Study of ASP1517 in Healthy Non-elderly Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Director, Astellas Pharma , Inc
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 1517-CL-0201
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; Safety and tolerability; Plasma concentration; ASP1517; FG-4592
MeSH Terms: interventions — roxadustat

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Experimental): single administration
  Interventions: Drug: ASP1517; Drug: Placebo
- Part 2 (Experimental): multiple administration
  Interventions: Drug: ASP1517; Drug: Placebo

INTERVENTIONS:
Drug: ASP1517 — oral
  Other Names: FG-4592
Drug: Placebo — oral

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of ASP1517 after single or multiple oral administration in healthy non-elderly adult male subjects.

DETAILED DESCRIPTION:
The study consists of two parts, single and multiple dose. Within each part participants will be randomized to either ASP1517 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Body weight: ≥50.0 kg, <80.0 kg
* BMI: ≥18.5 kg/m2, <25.0 kg/m2
* Eligible, as judged by the investigator/subinvestigator based on the results of physical examinations (subjective symptoms and objective findings) and all tests obtained at screening and up to the timing immediately before study medication
* Supine blood pressure: Systolic blood pressure ≥90 mmHg, ≤130 mmHg; Diastolic blood pressure ≤85 mmHg
* Pulse rate at rest in supine position: ≥40 bpm, <100 bpm

Exclusion Criteria:

* Received any investigational drugs in other clinical or post-marketing studies within 120 days before the screening assessment
* Donated 400 mL of whole blood within 90 days, 200 mL of whole blood within 30 days, or blood components within 14 days before the screening assessment
* Received medication within 7 days before hospital admission or is scheduled to receive medication
* History of drug allergies
* Upper gastrointestinal disease (e.g. nausea, vomiting, stomachache) within 7 days before the study
* Excessive smoking or drinking habit (measure of "excessive": alcohol: 45 g/day, smoking: 20 cigarettes/day)

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ASP1517 | During 2 weeks

SECONDARY OUTCOMES:
Pharmacokinetics of ASP1517 | During 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Kantou, Japan